CLINICAL TRIAL: NCT06307808
Title: Viral Immunity in TrAnsplanted Patients Depending on iMmunosupressIon
Brief Title: Viral Immunity in Solid Organ Transplant Recipients: Monitoring Of The Response To Hepatitis B Booster Vaccination
Acronym: VITAMIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other)
Responsible Party: Sponsor
Other Study IDs: Vitamin
Record Dates: First submitted 2023-11-27; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-09

CONDITIONS: HBV; Kidney Transplantation; Liver Transplantation
Keywords: Hepatitis B virus; Kidney transplantation; Liver transplantation; Tacrolimus; Belatacept; HBV
MeSH Terms: conditions — Hepatitis B | interventions — Tacrolimus; Calcineurin Inhibitors; Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells, plasma samples, whole blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Kidney transplant recipients, tacrolimus treated: Prevalent kidney transplant recipients, receiving tacrolimus as main immunosuppresant
  Interventions: Drug: Tacrolimus
- Liver transplant recipients, tacrolimus treated: Prevalent liver transplant recipients, receiving tacrolimus as main immunosuppressant
  Interventions: Drug: Tacrolimus
- Kidney transplant recipients, belatacept treated: Prevalent kidney transplant recipients, receiving belatacept as main immunosuppressant
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Tacrolimus — Immunosuppressive drug: main immunosuppressant is a calcineurin inhibitor (CNI), namely tacrolimus
  Other Names: Calcineurin inhibitor
  Groups: Kidney transplant recipients, tacrolimus treated; Liver transplant recipients, tacrolimus treated
Drug: Belatacept — Immunosuppressive drug: main immunosuppressant is a costimulation inhibitor, namely belatacept
  Other Names: Costimulation inhibitor; CTLA4-Ig
  Groups: Kidney transplant recipients, belatacept treated

SUMMARY:
Solid Organ Transplantation (SOT) is made possible by the use of a lifelong immunosuppressive treatment. This treatment limits the response of the immune system, enabling long-term survival of the transplanted organ, but also leading to weaker anti-infectious responses.

In this study, we will compare the response to a booster Hepatitis B vaccination (HBV) in SOT patients, either after kidney or liver transplantation. We will also compare the immune response depending on the immunosuppressive treatment.

In order to provide a detailed picture of the immune response, we will investigate the usual serological response (anti-HBs antibodies), but also the cellular memory (both T and B) using ELISpot assays and flow-cytometry, over a 6 months period following booster vaccination.

DETAILED DESCRIPTION:
Solid Organ Transplantation (SOT) is the reference treatment for end stage kidney disease (Kidney Transplantation, KT) and liver failure (Liver Transplantation, LT). As of 2023, an immunosuppressive treatment remains mandatory for long-term graft survival. This treatment translates into a weaker response to vaccines. The recent example of Severe Acute Respiratory Syndrom (SARS) - Coronavirus (CoV), SARS-CoV-2, showed different vaccinal responses depending on the immunosuppressive drug, comparing belatacept- to tacrolimus-based immunosuppression.

Hepatitis B virus (HBV)-vaccination is recommended in chronic kidney failure and liver failure. However, post-transplantation, a loss of HBV seroprotection is seen in ~ 30 % of the patients. A booster HBV vaccine dose is recommended in such case, but the evaluation of the response to this booster dose is limited.

In the Viral Immunity in TrAnsplanted patients depending on iMmunosupressIoN (VITAMIN) study, investigators will investigate the effect of a HBV-vaccine booster on the immune system, comparing KT recipients treated with Belatacept with KT and LT recipients treated with Tacrolimus. The VITAMIN study is a prospective observational study recruiting KT and LT recipients from the time of a booster HBV vaccine injection and over the following 6 months. The idea is to take advantage of this very particular sensitizing event, at a defined timepoint, to investigate the immune response to HBV through vaccination. Investigators will focus on comparing the immunological state before and after vaccination, in kidney and liver transplant recipients receiving immunosuppression.

The immunological state will be described through 1/ the antibody response, 2/ its phenotype (both exploring the T cell compartment and the B cell compartment, including memory B cells, using flow cytometry) and 3/ its functional response (through the ELISpot assessment of the T response against HBV HBs antigen). Sequential blood samples will be taken, using Peripheral Blood Monocytic Cells (PBMC). Also, investigators will focus on HBV-specific memory B cells, to detect potential antibody secreting cells. This project will provide a longitudinal picture of all immune compartments stimulated by HBV vaccination. This longitudinal picture will be compared between tacrolimus-treated KT and LT recipients and belatacept-treated KT recipients.

The main objective is to compare the serological response (anti-HBs antibodies) between tacrolimus- and belatacept-treated patients. The secondary objective is to describe and compare the phenotype and functional T and B responses between tacrolimus- and belatacept-treated patients.

Comparing different immunosuppressive regimen through the immunological responses, investigators aim at improving the personalization of the immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Kidney or liver transplant recipients
* Grenoble University Hospital regular follow-up
* Tacrolimus or belatacept treated
* Clinical indication for HBV booster vaccination

Exclusion Criteria:

* Pregnancy or lactating woman
* History of HBV infection (either anti-Hepatitis B capside antigen (HBc), positivity or HBV-DNA positivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having received a kidney or liver transplant, with a regular follow-up at Grenoble University Hospital. Patients should have received a previous HBV vaccination. Anti-HBs antibody titer should have decreased to < 10 mUI/ml or have decreased > 50 mUI/ml when compared to a pre-transplantion status.
  Patients should receive a tacrolimus or belatacept-based immunosuppression.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Titer of anti-HBs ELISA antibody | From enrollment to 6 months after inclusion
  Anti-HBs HBV serological response

SECONDARY OUTCOMES:
Number of anti-HBs memory B cells | From enrollment to 6 months post-enrollment
  B-ELISpot anti-HBs memory B cells

CONTACTS AND LOCATIONS:
Overall Officials: Thomas JOUVE, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, AURA, France

IPD SHARING:
Plan to Share IPD: Yes
Patients demographics and longitudinal HBV serological status
Supporting Information: Study Protocol, CSR
Time Frame: From study completion (expected 09/2025), for 5 years
Access Criteria: Researchers wishing to investigate with our data set will contact the primary investigator and discuss the research project.